CLINICAL TRIAL: NCT00023855
Title: A Phase I and Pharmacodynamic Study of Proteasome Inhibitor, PS-341, in Combination With Doxorubicin in Patients With Advanced Solid Tumors
Brief Title: PS-341 and Doxorubicin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068870; P30CA014520 (NIH); WCCC-CO-01901; NCI-3771
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2015-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Bortezomib; Doxorubicin

INTERVENTIONS:
Drug: bortezomib
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of combining PS-341 and doxorubicin in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of PS-341 in combination with doxorubicin in patients with advanced solid tumors.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of PS-341.

Patients receive PS-341 IV over 3-5 seconds on days 1, 4, 8, and 11; and doxorubicin IV on over 3-5 minutes on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of PS-341 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3-31 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor for which no curative treatment exists
* Measurable or evaluable disease
* No brain metastases or primary brain tumors

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* MUGA at least 45%

Other:

* No serious active infection
* No pre-existing neuropathy grade 2 or greater
* No other concurrent illness that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No prior cumulative dose of doxorubicin exceeding 280 mg/m^2

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent investigational or commercial agents for treatment of this malignancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P. Thomas, MD, PhD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] LoConte NK, Thomas JP, Alberti D, Heideman J, Binger K, Marnocha R, Utecht K, Geiger P, Eickhoff J, Wilding G, Kolesar J. A phase I pharmacodynamic trial of bortezomib in combination with doxorubicin in patients with advanced cancer. Cancer Chemother Pharmacol. 2008 Dec;63(1):109-15. doi: 10.1007/s00280-008-0719-5. Epub 2008 Mar 6. PMID 18322686